CLINICAL TRIAL: NCT03555019
Title: Effects of Nutrition Therapy on Growth, Inflammation and Metabolism in Immature Infants; a Double-blind Randomized, Controlled Trial
Brief Title: Nutrition Therapy in the Immature Infant (ImNuT)
Acronym: ImNuT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Umeå University (Other); University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Sissel Jennifer Moltu, MD, PhD, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2016-003700-31
Record Dates: First submitted 2018-04-10; First posted 2018-06-13 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Immature Infant; Essential Fatty Acid Deficiency
Keywords: Brain maturation; Postnatal growth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized-controlled. Parallel group, single center trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formulaid (Experimental): The intervention group will receive enteral supplementation with Formulaid containing ARA and DHA at a ratio of 2:1, from birth until 36 weeks PMA
  Interventions: Dietary Supplement: Formulaid
- MCT-oil (Active Comparator): The control group will receive enteral supplementation with MCT oil containing coconut and/or palm kern oil, from birth until 36 weeks PMA
  Interventions: Dietary Supplement: MCT-oil

INTERVENTIONS:
Dietary Supplement: Formulaid — Supplementation with ARA and DHA
  Arms: Formulaid
Dietary Supplement: MCT-oil — Supplementation with medium chain fatty acids
  Arms: MCT-oil

SUMMARY:
The primary objective of this double-blind randomized study is to assess the effects of an early, enhanced supply of the essential fatty acids (FAs) arachidonic acid (ARA) and docosahexaenoic acid (DHA) on brain maturation, clinical outcomes and quality of growth in immature infants (gestational age <29 weeks) as compared to standard nutrient supply.

DETAILED DESCRIPTION:
This is a double-blind randomized study. 172 preterm infants with gestational age < 29 weeks will be enrolled. The intervention group will receive enteral supplementation with essential fatty acids, arachidonic acid (ARA) and docosahexaenoic acid (DHA). The control group will receive standard supplementation with medium-chain triglycerides (MCT-oil). The main hypothesis is that early, enhanced supply of ARA and DHA will improve brain growth and maturation, as compared to standard nutrient supply. Secondary hypotheses are that early, enhanced supply of ARA and DHA will improve quality of growth and cognitive development as well as reduce the frequency of inflammation-related neonatal comorbidities and long-term cardiovascular disease risk. Primary endpoint will be assessed by magnetic resonance imaging (MRI) of the brain at term equivalent age.

ELIGIBILITY:
Inclusion Criteria:

* Extremely preterm infants born at Oslo University Hospital (OUH)
* Gestational age (GA) < 29 weeks
* Less than 48 hours of age at inclusion
* Signed informed consent and expected Cooperation of the patients for the treatment and follow up must be obtained and documented according to good clinical practice (GCP) and national/local regulations

Exclusion Criteria:

* Major congenital malformations which will affect growth and development
* Chromosomal abnormalities and other genetic diseases
* Critical illness with short life expectancy as defined by the study physician

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Brain maturation assessed by magnetic resonance imaging (MRI) | 40 weeks postmenstrual age (PMA)
  MRI with spectroscopy (MRS) and diffusion tensor imaging (DTI) will be used to examine myelinisation and quantification of anatomical structures as well as neuronal integrity and inflammation

SECONDARY OUTCOMES:
Weight gain | Weight will be recorded until 36 weeks PMA and at 3, 6, 12 and 24 months and 8 years corrected age.
  Weight measurements, including weight nadir.
Growth | Length and HC will be recorded until 36 weeks PMA and at 3, 6, 12 and 24 months and 8 years corrected age.
  Length and head circumference (HC).
Body composition | At 36 weeks PMA, 3 months and 2 years corrected age
  Body composition will be assessed using PEA POD, an air displacement plethysmography system and Dexa Scan.
Neonatal morbidities associated with inflammation | From birth til 36 weeks PMA
  Bronchopulmonary dysplasia (BPD), retinopathy of prematurity (ROP), necrotizing enterocolitis (NEC), white matter injury (WMI) of the brain, and late onset septicemia
Cerebral Background Activity evaluated by Electroencephalogram (EEG) | First week of life, 36 weeks PMA and 2 years corrected age (CA)
  EEG maturational changes will be examined as a function of time and as a function of gestational age
Neurodevelopment assessed by standardized motor and cognitive tests | 2 years corrected age (CA)
  Evaluation of psychomotor development by performing Bayley III and a standardized neurological examination
Lung function evaluated by tidal breathing measurements | 36 weeks PMA, 3 months and 2 years CA
  Tidal breathing measurements include tidal volume, respiratory rate, minute ventilation and fraction of expiratory time to peak tidal expiratory flow to total expiratory time
Cardiovascular Health assessed by echocardiography | First week of life, 2nd week of life, at 36 weeks PMA and 2 years CA
  Echocardiography will be used to follow the transition from fetal to completed neonatal circulation, to measure superior vena cava flow, and to study mycardial function by the use of conventional two-dimensional echocardiography and tissue Doppler imaging.
Blood pressure | First week of life and at 36 weeks PMA and 2 years CA
  Measurements of systolic, diastolic and mean pressure
Fatty acid (FA) profiles in blood | From birth until 36 weeks PMA
  Repeated dried blood spots (DBS) samples with approximately 10 µL blood will be collected for FA analyses. These analyses are important for assessing efficacy and protocol compliance. We will also collect 10 µL of fullblood for assessment of total lipid profile (Lipidomics).
Markers of inflammation | From birth until 36 weeks PMA
  Inflammation panels will be used to assess markers of inflammation in fullblood and sputum
Markers of metabolic status | From birth until 36 weeks PMA
  Metabolic pathway analyses (http://omictools.com/metabolic-pathways-category) will be performed to analyse and describe the metabolic conditions of the infants during hospitalization. Metabolites outside the standard clinical chemistry parameters will also be investigated ("untargeted metabolomics). Metabolomics will be performed by the use of dried blood spot samples
Markers of nutritional status in blood | From birth until 36 weeks PMA
  The concentrations of electrolytes, minerals, albumin, alkaline phosphatase, vitamin A and D will be assessed regularly during hospitalization
Micronutrient content in urine | From birth until 36 weeks PMA
  Spot urine will be obtained regularly to study the changes in electrolyte- and mineral homeostasis during the first week of life as well as during the phase of steady growth
Evaluation of nutrient composition of expressed breast milk | From birth until 36 weeks PMA
  Repeated samples of breast milk will be collected for FA analyses, macronutrient content and vitamin A
Gut microbiota | From birth until 36 weeks PMA
  Repeated samples of feces will be used to study the early fecal microbiota
Inflammatory markers in sputum | From birth until 36 weeks PMA
  We will analyze the Expression of a standardized panel of inflammatory markers in collected laryngeal or tracheal secretion

CONTACTS AND LOCATIONS:
Overall Officials: Tom Stiris, MD, ass prof, Study Director — Departement of Neonatal Intensive care, Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 6 months of study completion

REFERENCES:
- [Derived] Gunnarsdottir G, Rossholt ME, Nordvik T, Wendel K, Aas MF, Skarbo AB, Aulie VS, Stiris T, Ramm-Pettersen A, Pfeiffer HC, Moltu SJ. High dose arachidonic and docosahexaenoic acid in very preterm infants and neurodevelopment at 2 years - A double-blind randomized controlled trial. Clin Nutr. 2025 Aug;51:198-205. doi: 10.1016/j.clnu.2025.05.019. Epub 2025 Jun 4. PMID 40580806
- [Derived] Moltu SJ, Nordvik T, Rossholt ME, Wendel K, Chawla M, Server A, Gunnarsdottir G, Pripp AH, Domellof M, Bratlie M, Aas M, Huppi PS, Lapillonne A, Beyer MK, Stiris T, Maximov II, Geier O, Pfeiffer H. Arachidonic and docosahexaenoic acid supplementation and brain maturation in preterm infants; a double blind RCT. Clin Nutr. 2024 Jan;43(1):176-186. doi: 10.1016/j.clnu.2023.11.037. Epub 2023 Nov 29. PMID 38061271
- [Derived] Rossholt ME, Bratlie M, Wendel K, Aas MF, Gunnarsdottir G, Fugelseth D, Pripp AH, Domellof M, Stordal K, Stiris T, Moltu SJ. Effect of arachidonic and docosahexaenoic acid supplementation on quality of growth in preterm infants: A secondary analysis of a randomized controlled trial. Clin Nutr. 2023 Dec;42(12):2311-2319. doi: 10.1016/j.clnu.2023.10.005. Epub 2023 Oct 17. PMID 37856920
- [Derived] Wendel K, Aas MF, Gunnarsdottir G, Rossholt ME, Bratlie M, Nordvik T, Landsend ECS, Fugelseth D, Domellof M, Pripp AH, Stiris T, Moltu SJ. Effect of arachidonic and docosahexaenoic acid supplementation on respiratory outcomes and neonatal morbidities in preterm infants. Clin Nutr. 2023 Jan;42(1):22-28. doi: 10.1016/j.clnu.2022.11.012. Epub 2022 Nov 17. PMID 36473425
- [Derived] Hortensius LM, Hellstrom W, Savman K, Heckemann RA, Bjorkman-Burtscher IM, Groenendaal F, Andersson MX, Nilsson AK, Tataranno ML, van Elburg RM, Hellstrom A, Benders MJNL. Serum docosahexaenoic acid levels are associated with brain volumes in extremely preterm born infants. Pediatr Res. 2021 Dec;90(6):1177-1185. doi: 10.1038/s41390-021-01645-w. Epub 2021 Aug 14. PMID 34392310
- [Derived] Wendel K, Pfeiffer HCV, Fugelseth DM, Nestaas E, Domellof M, Skalhegg BS, Elgstoen KBP, Rootwelt H, Pettersen RD, Pripp AH, Stiris T, Moltu SJ; ImNuT Collaboration Group. Effects of nutrition therapy on growth, inflammation and metabolism in immature infants: a study protocol of a double-blind randomized controlled trial (ImNuT). BMC Pediatr. 2021 Jan 7;21(1):19. doi: 10.1186/s12887-020-02425-x. PMID 33407269